CLINICAL TRIAL: NCT04134923
Title: Imaging Biomarkers in Preclinical and Symptomatic AD. (ACS PiB IND)
Brief Title: Imaging Biomarkers in Preclinical and Symptomatic AD
Acronym: ACS_PIB_IND
Status: Recruiting | Type: Observational
Sponsor: Tammie L. S. Benzinger, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Tammie L. S. Benzinger, MD, PhD, Professor of Radiology, Neuroradiology Section Professor of Neurological Surgery Director, Knight Alzheimer Research Imaging Program, Washington University School of Medicine
Organization: Washington University School of Medicine (Other)
Other Study IDs: 201906028
Record Dates: First submitted 2019-10-18; First posted 2019-10-22 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's disease; neurology; radiology; Nuclear medicine
MeSH Terms: conditions — Alzheimer Disease | interventions — 2-(4'-(methylamino)phenyl)-6-hydroxybenzothiazole

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- [11C] Pittsburgh Compound-B (PIB): Using [11C] Pittsburgh Compound-B (PIB) to look for biomarkers in preclinical and symptomatic AD.
  Interventions: Drug: [11C] Pittsburgh Compound-B (PIB)

INTERVENTIONS:
Drug: [11C] Pittsburgh Compound-B (PIB) — Participants will receive a single intravenous bolus injection of 6.0 - 20.0 mCi (222-740 MBq) of the investigational radiotracer [11C] PIB. Participants will then undergo a [11C] PIB PET/CT scan conducted in the Center for Clinical Imaging Research (CCIR) facility.

SUMMARY:
The purpose of this research study is to evaluate adult children of parents with and without Alzheimer's disease which represent an ideal population for investigating the biological changes that precede the clinical onset of AD. The investigators will be imaging the brain to detect the presence of amyloid deposits (plaques in the brain). Amyloid is a protein that may be related to dementia of Alzheimer's disease (DAT).

DETAILED DESCRIPTION:
This study will use a radioactive tracer called [11C]-Pittsburgh Compound B (11C]PIB), which is a tracer that binds to beta amyloid protein in the brain. This compound is considered investigational, which means that it has not been approved by the United States Food and Drug Administration (FDA).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, any race;
* Age ≥ 18 years;
* Active participants currently enrolled in the Knight Alzheimer's Disease Research Center (ADRC) at Washington University.

Exclusion Criteria:

* Hypersensitivity to [11C] PIB or any of its excipients;
* Contraindications to PET, CT or MRI (e.g. electronic medical devices, inability to lie still for extended periods) that make it unsafe for the individual to participate;
* Severe claustrophobia;
* Women who are pregnant or breast-feeding will be excluded from PIB PET participation;
* Has any condition that, in the opinion of the Sponsor-Investigator or designee could increase risk to the subject, limit the subject's ability to tolerate the research procedures, or interfere with collection of the data;
* Currently participating in any clinical trial which involves an active study medication or placebo within the past 30 days before scanning and up to 2-weeks past the imaging visit.
* Current or recent (within 12 months prior to screening) participation in research studies involving radioactive agents such that the total research-related radiation dose to the participant in any given year would exceed the limits set forth in the U.S. Code of Federal Regulations (CFR) Title 21 Section 361.1. https://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfcfr/CFRSearch.cfm?FR=361.1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Active participants currently enrolled in the Knight Alzheimer's Disease Research Center (ADRC) at Washington University.
Sampling Method: Non-Probability Sample
Enrollment: 375 (Estimated)
Dates: Start 2021-06-08 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
develop an integrated timeline for the imaging changes which occur during the transition from asymptomatic to symptomatic AD | 5 years
  the annual rate of CDR progression will accelerate due to the aging of the ACS cohort., and estimate that among ~375 ACS participants who either remain CDR 0 currently and will continue to be clinically assessed or will be the new future enrollees, a total of 45 individuals will progress to CDR>0 by the end of next funding cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Tammie Benzinger, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No